CLINICAL TRIAL: NCT06344221
Title: Post-stroke Haptic Feedback Use Deficit: A Comparative and Reliability Study
Acronym: HapticS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Paris Brain Institute (ICM) (Other); Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A00954-41
Record Dates: First submitted 2024-02-16; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Upper Extremity Paresis; Manual Dexterity; Sensory Integration Dysfunction; Vibration; Disorder
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young Healthy Controls (Active Comparator): The 3 groups, made up of participants with different pathologies and ages, will receive the same intervention (clinical motor and sensory tests and optional TMS). We are studying the difference in results between these groups.
  Interventions: Device: Dextrain Manipulandum and haptic feedback device
- Healthy controls matched in age and sex with stroke patients (Active Comparator): The 3 groups, made up of participants with different pathologies and ages, will receive the same intervention (clinical motor and sensory tests and optional TMS). We are studying the difference in results between these groups.
  Interventions: Device: Dextrain Manipulandum and haptic feedback device
- Chronic stroke patients (Experimental): The 3 groups, made up of participants with different pathologies and ages, will receive the same intervention (clinical motor and sensory tests and optional TMS). We are studying the difference in results between these groups.
  Interventions: Device: Dextrain Manipulandum and haptic feedback device

INTERVENTIONS:
Device: Dextrain Manipulandum and haptic feedback device — Assessment of key components of manual dexterity in addition to vibrotactile stimulation on the fingers and wrist.
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
The aim of this comparative and reliability study is to highlight a deficit in the use of vibrotactile sensory feedback (haptic effect) in the planning and execution of fine manual dexterity movements after stroke. The investigators will include 3 groups of subjects, 1 group of young healthy subjects, 1 of older subjects matched in age and sex to the group of chronic stroke patients. Participants will take part in clinical tests of fine motor skills and sensitivity and will use a device to assess the key components of manual dexterity, to which vibrotactile sensors will be added. If they so wish, participants will be able to take part in a transcranial magnetic stimulation (TMS) study to assess the facilitation of cortical excitability due to the haptic effect.

DETAILED DESCRIPTION:
Firstly, the investigators would like to carry out a study into the validity of measuring haptic deficits using vibro-tactile sensors positioned on the hands of chronic stroke patients and young and elderly healthy subjects. They believe that identifying the haptic deficit using a simple and rapid method, in combination with motor training, could make it possible to improve the prediction of recovery and personalise the rehabilitation of manual dexterity deficits after stroke. They will also compare the effect of tactile feedback with that of auditory feedback in order to study the specificity of the effect of this feedback on manual dexterity. In the second part, to better understand this and to study the cortical mechanisms involved in sensory-motor integration, the investigators propose to measure the haptic effect on cortical excitability in stroke patients and healthy subjects using Transcranial Magnetic Stimulation (TMS).

ELIGIBILITY:
Inclusion Criteria for healthy controls:

* between 18 and 40 years old
* or age and sex match with chronic stroke patients
* Ability to perform motor, cognitive (MOCA score ≥26/30) and sensory assessment

Inclusion Criteria for chronic stroke patients:

* More than 18 years old
* Ability to perform motor, cognitive (MOCA score ≥26/30) and sensory assessment
* First symptomatic stroke more than 6 months ago
* Upper limb paresis (≤4/5 on the MRC scale)
* Feel ≥3/6 touch on the index and thumb fingers
* Box and Blocks test score between 1 and 54 blocks / min

Exclusion Criteria:

* Contraindication to TMS (epilepsy, metal implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Assessing haptic effect during a dexterity exercise with and without sensory feedback: finger independence | 1 day
  Comparison of finger independence, assessed with the Dextrain Manipulandum tool with and without sensory feedback (vibrations on the fingers). Measurement of the difference in motor performance between the condition with and without vibrations.

SECONDARY OUTCOMES:
Assessing haptic effect during another dexterity exercise with and without sensory feedback: the force control of the index | 1 day
  Comparison of finger force control, assessed with the dextrain manipulandum tool with and without sensory feedback (vibrations on the fingers). Measurement of the difference in motor performance between the condition with and without vibrations.
Assessing haptic effect during another dexterity exercise with and without sensory feedback: the rhythm capacity | 1 day
  Comparison of rhythm capacity, assess with the dextrain manipulandum tool with and without sensory feedback (vibrations on the fingers). Measurement of the difference in motor performance between the condition with and without vibrations.
Correlation between clinical assessment and haptic measure | 1 day
  Research the link between haptic feedback deficits and motor disorders of manual dexterity
Assessment of the feasibility of the haptic measures | 1 day
  Assessment of Intrinsic motivation survey to quantify the feasibility of the haptic device. The score will be from 0 to 7, 7 meaning an excellent motivation of the patient to use the device
Assessment of the benefits of the haptic measures | 1 day
  Assessment of User Engagement scale to quantify the benefits perceived by the subject in relation to the haptic device. The score will be from 0 to 10, 10 meaning an excellent interest of the patient for the device
Study the test re-test reliability of the haptic device by comparing the haptic effect on dexterity assessed at the beginning and end of the session by the same evaluator | 1 day
  The same examinator will assess haptic effect at the beginning and at the end of the session
Assessment of the impact of age on the dexterity performances (Finger independence, force control of the index and rhythm capacity) | 1 day
  Comparison of the haptic effect (difference in motor performance between the conditions with and without vibrations on the fingers) between the groups of young healthy subjects and the group of healthy subjects of comparable age and sex to chronic stroke patients
Measurement of the manual dexterity facilitation between tactile (haptic device with vibrations on the fingers) and auditory feedback (sounds during the dexterity tasks) | 1 day
  To compare the effect of tactile (vibrations on the fingers during dexterity assessments) modality facilitation versus auditory feedback on dexterity (finger independence, force control of the index and rhythm capacity) in stroke patients, young healthy subjects and healthy subjects of comparable age and sex to chronic stroke patients
Transcranial magnetic stimulation (TMS) | 1 day
  Difference in cortical excitability in the anticipatory phase of force generation with the index finger between conditions without and with vibro-tactile stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Turc, Principal Investigator — GHU Psychiatrie et Neurosciences de Paris

IPD SHARING:
Plan to Share IPD: No